CLINICAL TRIAL: NCT04277793
Title: Feasibility Evaluation of a Monitored Self-guided Digital Cognitive Behavioural Therapy Format: an Uncontrolled Trial of a Problem Solving Intervention for Depression and Anxiety
Brief Title: Feasibility Evaluation of a Monitored Self-guided Cognitive Behavioural Therapy Digital Format
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Martin Kraepelien, Licensed clinical psychologist, Principal investigator, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVPSY290/19
Record Dates: First submitted 2020-02-11; First posted 2020-02-20 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Depressive Symptoms; Anxiety
Keywords: CBT; Digital; Internet-based; Depression; Anxiety; Self-guided; Problem Solving; ICBT
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitored self-guided problem solving intervention (Experimental): Monitored self-guided problem solving intervention
  Interventions: Behavioral: Monitored self-guided problem solving

INTERVENTIONS:
Behavioral: Monitored self-guided problem solving — Problem Solving is a behavioral modification intervention focusing on the training of adaptive problem-solving skills in order to cope more effectively with everyday stressful events.

SUMMARY:
The purpose of the study is to evaluate the feasibility of a new monitored self-guided digital cognitive behavioural therapy format through one of the key components of an intervention for depression and anxiety (Problem Solving) and to answer the question: Do patients with significant levels of depression and/or anxiety symptoms consider the monitored self-guided digital format usable and credible? An uncontrolled trial will explore participant's usability and treatment credibility ratings.

DETAILED DESCRIPTION:
Objective. The purpose of the study is to evaluate the feasibility of a new monitored self-guided digital cognitive behavioural therapy format through one of the key components of an intervention for depression and anxiety (Problem Solving) and to answer the question: Do patients with significant levels of depression and/or anxiety symptoms consider the monitored self-guided digital format usable and credible?

Background. Problem Solving is a behavioral modification intervention focusing on the training of adaptive problem-solving skills in order to cope more effectively with everyday stressful events. It is one of the most well-examined therapeutic interventions for depression, with reliable support regarding symptom improvement in depression traditionally delivered with therapist-guidance when administered via the Internet. Since a new monitored self-guided digital intervention for depression and anxiety has been developed, including the key component Problem Solving, it is of importance to assess both the usability and treatment-credibility of this format to evaluate if it is feasible.

Methodology. Based on similar feasibility studies including around ten participants, a number of 16-30 participants will be included in this study to compensate for potential drop-outs. Participants will be recruited via a psychiatric clinic belonging to Stockholm County Council in Stockholm, Sweden, and will be patients in queue for treatment for depression and/or anxiety in a psychiatric setting. Inclusion criteria will be significant depression and/or anxiety symptoms. The participants included in the study will access the key component Problem Solving during four weeks while being on waitlist for regular treatment. They will be introduced to the intervention as a self-explanatory tool with possible beneficial effects on depression symptoms. Self-assessments will be carried out during the intervention. The scores on these scales will be compared to available published data from these scales from evaluations of therapist-guided Internet-based interventions if available, and otherwise data from these scales from studies on other digital interventions for mental health. The participants will also answer questions concerning their experience of the format.

ELIGIBILITY:
Inclusion Criteria:

Significant depression and/or anxiety symptoms measured with Patient Health Questionnaire (PHQ-9) and General Anxiety Disorder (GAD-7) (i.e. a PHQ-9 and/or GAD-7 score of ≥5).

Exclusion Criteria:

1. insufficient Swedish knowledge
2. minor (i.e. age <18 years)
3. high suicide risk (i.e. a score ≥4 on the ninth item on the Montgomery Åsberg Depression Scale, MADRS-S)
4. lack of access to a device with Internet connection (e.g. computer, mobile, tablet)
5. lack of access to a phone on which calls and SMS can be received
6. psychiatric or somatic problems that must be prioritized before or become an excessive obstacle to the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | immediately after the intervention
  Self-rated assessment of usability, higher score is better
Treatment Credibility Scale | immediately after the intervention
  Self-rated assessment of treatment credibility, higher score is better

SECONDARY OUTCOMES:
Negative Effects Questionnaire | immediately after the intervention
  Self-rated assessment of negative treatment effects, lower score is better
Negative Effects Questionnaire | During the intervention: 2 weeks from baseline
  Self-rated assessment of negative treatment effects, lower score is better
Patient Health Questionnaire - 9 | Change from baseline immediately after the intervention
  Self-rated depressive symptoms, lower score is better
Generalized Anxiety Disorder - 7 | Change from baseline immediately after the intervention
  Self-rated anxiety symptoms, lower score is better
System Usability Scale | During the intervention: 2 weeks from baseline
  Self-rated assessment of usability, higher score is better
Treatment Credibility Scale | During the intervention: 2 weeks from baseline
  Self-rated assessment of treatment credibility, higher score is better

OTHER OUTCOMES:
Evaluation of treatment format | During the intervention: 2 weeks from baseline
  Written quantitative and qualitative questions concerning the treatment format
Evaluation of treatment format | immediately after the intervention
  Written quantitative and qualitative questions concerning the treatment format
Interview concerning treatment format | immediately after the intervention
  Phone interview with qualitative questions concerning the treatment format

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum för Psykiatriforskning, Stockholm, Sweden